CLINICAL TRIAL: NCT05940077
Title: Influence of Community-based Group Exercise on Fall Risk in Parkinson's Disease
Brief Title: Community Exercise for Fall Risk in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Idaho State University (Other)
Responsible Party: Principal Investigator, Evan Papa, Associate Professor, Idaho State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2019-205; 5U54GM104944-08 (NIH)
Record Dates: First submitted 2023-06-27; First posted 2023-07-11 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease; Fall; Exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community-based exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Community-based exercise involving non-contact boxing and individualized balance training

SUMMARY:
Parkinson's disease (PD) affects approximately 1 million people in the United States and causes significant fall risks. This study aims to develop a community-based exercise program that reduces falls in persons with PD. By combining individualized balance activities with group boxing training, the study seeks to identify modifiable risk factors, improve balance dysfunction, and reduce falls. The findings will inform clinical practice, offering a community-based exercise model to address the urgent need for effective fall prevention interventions in PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disorder and effects approximately 1 million people in the United States. Falls are a significant problem for persons with PD, with incidence rates ranging from 37-80% each year. The long-term goal of this research is to develop exercise training programs to reduce falls in persons with PD.

Physical activity and exercise are commonly understood to provide significant benefits in functional mobility for persons with PD. Unfortunately, the translation of improved mobility to an actual reduction in falls has been recalcitrant to traditional exercise therapies. The following proposal is aimed at identifying the modifiable risk factors for falls in persons with PD and characterizing the effect of a novel exercise intervention on fall risk. The investigators will conduct a 12 week community-based exercise program in 20 individuals in which two validated forms of exercise training will be combined into one program. Specifically, individualized balance activities tailored to different domains of balance dysfunction for each individual will be combined with non-contact group boxing training to maximize the therapeutic benefit. The research aims of this investigation are 1) identify the individual characteristics of responders to exercise such as modifiable factors like lower-extremity kinematic joint range of motion and balance domain dysfunction at baseline, and 2) determine if a novel community-based exercise regimen that combines accepted balance and strength training protocols can synergistically improve balance dysfunction and reduce falls.

The benefits of exercise in general on PD are undisputed, but there remains an urgent, unmet need for the identification of exercise interventions that can reduce falls. The proposed research is significant because it is expected to provide evidence that a novel community-based exercise program is capable of improving functional mobility in such a way that it can reduce fall incidence for persons with PD. The research aims in this proposal are expected to directly inform clinical practice for rehabilitation providers by identifying the modifiable risk factors that lead to falls in PD and delivering a community-based exercise model that can reduce the harmful effects of falls in this population.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic PD; Male or female 30 years or older at time of PD diagnosis; Hoehn & Yahr (H&Y) stages 1.0-3.0; Ability to provide informed consent in accordance with Good Clinical Practice (GCP) and local regulations.

Exclusion Criteria:

* Idiopathic PD H&Y stage 4-5, in order to constrain motor dysfunctions to mild-to-moderate PD; Confirmed or suspected atypical parkinsonian syndromes due to drugs, metabolic disorders, encephalitis, or degenerative diseases; Presence of definite dementia by Montreal Cognitive Assessment (MoCA <21); Central or peripheral nervous system disorders (other than PD); Myopathic disease (e.g. focal myopathy) that affects skeletal muscle structure/function; Severe cardiovascular disease that limits exercise abilities.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Idaho State University, Pocatello, Idaho, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants may be excluded at this point if they demonstrate the presence of definite dementia, determined by Montreal Cognitive Assessment (MoCA < 21).
Period: Overall Study
Arm/Group | Community-based Exercise
Started | 20
Completed | 19
Not Completed | 1
Not completed — the presence of definite dementia, determined by Montreal Cognitive Assessment (MoCA < 21) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Community-based Exercise
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (4.6)
Hoehn & Yahr [Mean (Standard Deviation); unit: units on a scale] — The scale has been used for the staging of the functional disability associated with Parkinson's disease. It helps in describing the progression of the disease through various stages, thus allowing the measurement of the severity of the disease.
  Scale range = 1-5 (higher values = worse disease severity)
  units on a scale | 2.0 (0.7)
UPDRS (motor) [Mean (Standard Deviation); unit: units on a scale] — The Unified Parkinson's Disease Rating Scale (UPDRS) was developed to evaluate various aspects of Parkinson's disease (PD) including non-motor and motor experiences of daily living and motor complications. We are using the motor portion in this study. It characterizes the extent and burden of the motor complications of the disease (eg., postural instability, tremor, etc.).
  Scale = 0 - 108 (higher values = increase severity of disease)
  units on a scale | 16.9 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Falls Experienced During the Study Period as Reported by Self-report
Description: Higher scores = worse outcome
Time Frame: Baseline and Post-Intervention at approximately 12 weeks
Measure: Mean (Standard Error); unit: self-reported falls
Groups:
- Baseline; Post Intervention: Community-based exercise involving non-contact boxing and individualized balance training
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 20 | 20
self-reported falls | 16 (1.89) | 7 (0.83)

2. Secondary Outcome: TUG
Description: The "timed up and go test" (TUG) is a simple test of the subjects' ability to understand an instruction and perform the task of standing, walking 10ft, turning around, returning 10ft and sitting down Timed Up and Go, higher scores = worse outcome
Time Frame: Baseline and Post-Intervention at approximately 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 20 | 20
seconds | 11.02 (3.28) | 8.13 (1.74)

3. Secondary Outcome: BBS
Description: The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
  Scale = 0 - 56 (higher scores = better function)
Time Frame: Baseline and Post-Intervention at approximately 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 20 | 20
score on a scale | 40.47 (9.51) | 46.84 (6.73)

4. Secondary Outcome: ABC
Description: The Activities-Specific Balance Confidence (ABC) scale is a self-report measure of balance confidence in performing various activities without losing balance or experiencing a sense of unsteadiness. The ABC Scale has 16 questions that require the patient to rate his/her confidence that he/she will not lose balance or become unsteady while performing various activities.
  Scale: 0 - 100 (higher scores = better confidence)
Time Frame: Baseline and Post-Intervention at approximately 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 20 | 20
score on a scale | 78.92 (8.74) | 86.05 (9.45)

5. Secondary Outcome: 5-STS
Description: The Five Times Sit-to-Stand Test (5-STS) is used to asses functional lower extremity strength, transitional movements, balance, and fall risk in older adults. Scoring is based on the amount of time (to the nearest decimal in seconds) a patient is able to transfer from a seated to a standing position and back to sitting five times.
  Higher scores = Worse outcome
Time Frame: Baseline and Post-Intervention at approximately 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Baseline | Post Intervention
Number analyzed (Participants) | 20 | 20
seconds | 15.58 (3.39) | 11.53 (3.08)

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Arm/Group | Community-based Exercise
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT05940077/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT05940077/SAP_001.pdf
  • Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/77/NCT05940077/ICF_002.pdf